CLINICAL TRIAL: NCT05732363
Title: Evaluation of Different Methods to Measure Muscle Mass and Strength in a Population With Class II/III Obesity: A Follow-up Study
Brief Title: Evaluation of Different Methods to Measure Muscle Mass and Strength in a Population With Class II/III Obesity
Acronym: MUSCLE-II
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Dionne Sizoo, Senior researcher, Frisius Medisch Centrum
Other Study IDs: MCLeeuwarden
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-11

CONDITIONS: Obesity, Morbid
Keywords: Muscle mass; Sonography
MeSH Terms: conditions — Obesity, Morbid | interventions — Ultrasonography; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: The population will consist of patients, who have participated in the MUSCLE study and have received bariatric surgery at the CON / MCL. A potential subject who meets any of the following criteria will be excluded from participation in this study:
  * Inability to communicate in either Dutch or English
  * Weight over 204 kilograms (due to limitations of the DXA)
  * Pregnancy
  * Pacemaker
  Interventions: Device: Ultrasonography; Radiation: Dual-energy X-ray Absorptiometry

INTERVENTIONS:
Device: Ultrasonography — The US muscle measurement will be performed with the handheld portable Philips Lumify Sonography connected to a Samsung tablet. The measurement will take approximately 5-10 minutes. A seven-point measurement has to be performed based on the seven-site Jackson Pollock Generalized Prediction Equations for circumference and skinfold thickness measurements.6,7
  Other Names: ultrasound
Radiation: Dual-energy X-ray Absorptiometry — The brand of the DXA scanner is the Hologic Discovery A, which has a weight limit of 204 kilograms. During the DXA scan, patients will be exposed to radiation, which is approximately 0.2 micro Sievert (µSv) for measuring body composition. For comparison: the average amount of background radiation per hour is approximately 0.23 µSv. The DXA body composition scan will be performed according to standard protocol by a specialized technician.

SUMMARY:
Rationale: Weight loss therapies should aim to reduce fat mass while preserving both muscle mass and muscle strength. Consequently, there is a need for validated methods to measure muscle mass and strength. Current methods are either expensive and require trained technicians, or have not been validated in populations with class II/III obesity (BMI > 35 kg/m2). In our previous studies (MUST-MOP and MUSCLE study), we have validated the use of ultrasound (US) for the measurement of lean mass (a proxy for muscle mass) in a population with obesity. These studies showed that the use of US for the measurement of lean mass was feasible, reliable and valid. The aim of the current study is to validate the use of US for the measurement of lean mass after weight loss in a population of bariatric surgery patients.

Objective: Primary objective: To assess the validity of US to measure lean mass after weight loss in a population of bariatric surgery patients.

Secondary Objectives:

* To assess de differences in lean mass between DXA and US in this study compared to the MUSCLE-study.
* To assess how the lean mass has changed after bariatric surgery and the effects of lean mass on total weight loss and resolution of comorbidities
* To assess whether the change in lean mass has an effect on serum levels of markers for muscle mass.

Study design: This study is an observational follow-up study of the MUSCLE study and will take place in the Centre Obesity Northern-Netherlands (CON) at the Medical Centre Leeuwarden (MCL).

Study population: The population will consists of participants, who have participated in the MUSCLE study and have received bariatric surgery at the CON / MCL.

Main study parameters/endpoints: The main parameters of this study are: lean mass measured by DXA and US. The main endpoint of this study is the validity of the US measurement of lean mass compared to DXA.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no direct benefits for the participants. However, the results of this study can help to further validate the ultrasound as a cheaper and more accessible method to measure muscle mass. This can potentially be used in standard clinical care to assess muscle mass of patients during weight loss.

• The additional time investment: during first year follow-up appointment approximately 30 minutes.

The risks of most test are minor, even the small amount of radiation exposure, which means the risks and burden of this study outweigh the potentially obtainable knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Participation MUSCLE study
* ±1 year after bariatric surgery

Exclusion Criteria:

* Inability to communicate in either Dutch or English
* Weight over 204 kilograms (due to limitations of the DXA)
* Pregnancy
* Pacemaker

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients, who have participated in the MUSCLE study and have received bariatric surgery at the CON / MCL.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
lean mass measured by dual-energy X-ray absorptiometry | 1 time, 1 year after surgery
  gold standard
lean mass measured by ultrasound | 1 time, 1 year after surgery
  using LLM7 and LLM3 formulas

SECONDARY OUTCOMES:
weight loss after surgery | 1 time, 1 year after surgery
  total weight loss and excess weight loss (after bariatric surgery)
change in lean mass | 1 time, 1 year after surgery
  after bariatric surgery
comorbidity status | 1 time, 1 year after surgery
  Number of patients with resolution, improvement, same/worsened of comorbidities
blood parameters (e.g. CK, CRP, cystatin C, myoglobine) | 1 time, 1 year after surgery
  Concentration of blood parameters (e.g. CK, CRP, cystatin C, myoglobine)

CONTACTS AND LOCATIONS:
Overall Officials: Marloes Emous, PhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No